CLINICAL TRIAL: NCT04832568
Title: Perioperative EEG-Monitoring and Postoperative Delirium in Patients Undergoing Cardiovascular Surgery: a Prospective Observational Study
Brief Title: Perioperative EEG-Monitoring and Postoperative Delirium in Patients Undergoing Cardiovascular Surgery
Status: Recruiting | Type: Observational
Sponsor: Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Hua Zheng, Principal Investigator, Huazhong University of Science and Technology
Other Study IDs: TJMZK202101
Record Dates: First submitted 2021-03-31; First posted 2021-04-06 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Delirium
MeSH Terms: conditions — Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Delirium is determined by CAM or CAM-ICU score
- No delirium is determined by CAM or CAM-ICU score

SUMMARY:
Postoperative delirium is common in patients undergoing cardiovascular surgery and associated with poor outcomes. However the pathogenesis of postoperative delirium is poorly understood. Multichannel electroencephalogram is a recognized tool for identifying neurophysiologic states during anesthesia, sleep, and arousal. The aim of the current study is to evaluate the mechanisms and predictors of postoperative delirium in patients undergoing cardiovascular surgery using electroencephalogram.

ELIGIBILITY:
Inclusion Criteria:

1. age of at least 18 years
2. normal cognitive function at the time of enrollment evidenced by a Mini-Mental State Examination (MMSE) score of more than 24 of 30
3. Chinese Mandarin as the native language
4. providing informed consent

Exclusion Criteria:

1. pre-existing delirium assessed according to the Confusion Assessment Method (CAM)
2. history of neurological or psychiatric disease
3. impaired vision or auditory function which may effect the assessments
4. unwillingness to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing cardiovascular surgery
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-06-17 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of postoperative delirium | After surgery through to postoperative day 7
  The incidence of postoperative delirium was determined according to the Confusion Assessment Method (CAM) diagnostic algorithm. The algorithm consists of four clinical criteria: (1) acute onset and fluctuating course, (2) inattention, (3) disorganized thinking, and (4) altered level of consciousness. To define a patient as having delirium, both the first and the second criteria have to be present, as well as either the third or the fourth criteria. The CAM-ICU will be used for patients who are intubated in the postoperative period.

SECONDARY OUTCOMES:
Relative power of each brain waves | During the stay of the patient in the operating room, after surgery through to postoperative day 7
  Electroencephalogram data were acquired using a 32-channel electroencephalogram recording system (Brain Products, Germany). A 5 min, baseline, eyes-closed recording was conducted at the preoperative holding room when the patient was at rest. Recording of electroencephalogram was commenced before the start of anesthetic induction and was stopped before discharge of the patient from the operating room. We defied delta (1 to 3 Hz), theta (4 to 7 Hz), alpha (8 to 12 Hz), and beta (13 to 40 Hz) frequency bands. And then, the relative power of each frequency bands to the total power of the sum is calculated.
Duration of delirium | After surgery through to postoperative day 7
Severity of delirium | After surgery through to postoperative day 7
  Delirium severity is evaluated both as the peak (highest) and sum Confusion Assessment Method - Severity (CAM-S) score over all hospital days. The CAM-S includes two forms: a Short Form (CAM-S Short Form, based on the 4-item algorithm, the sum of score ranging from 0 to 7, with 7 being the most severe) and a Long Form (CAM-S Long Form, based on the 10-item CAM instrument, the sum of score ranging from 0 to 19, with 19 being the most severe).
Worst daily pain scores at rest | After surgery through to postoperative day 7
  Pain scores will be collected three times daily using a numeric rating scale (0, no pain, to 10, worst possible pain).
Worst daily pain scores with exertion (deep breathing and cough) | After surgery through to postoperative day 7
  Pain scores will be collected three times daily using a numeric rating scale (0, no pain, to 10, worst possible pain).
Length of stay in the Intensive Care Unit (ICU) | through study completion, an average of 5 days
  Measured in days admitted in the ICU
Length of hospital stay | through study completion, an average of 10 days
  Measured in days admitted in the hospital

OTHER OUTCOMES:
Biomarkers | before and after surgery in operating room, after surgery through to postoperative day 7
  Identify biomarkers (such as Ubiquitin carboxyl-terminal hydrolase L1 (UCH-L1), brain-derived neurotrophic factor (BDNF), and metalloproteases-9 (MMP-9) )of delirium and neural damage through changes in circulating plasma proteins and molecules

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anaesthesiology, Tongji Hospital of Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China